CLINICAL TRIAL: NCT01631058
Title: Immunosuppression in Renal Transplantation in The Elderly: Time to Rethink. - nEverOld Study
Brief Title: Renal Transplantation in the Elderly - nEverOld Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26423
Record Dates: First submitted 2012-06-21; First posted 2012-06-28 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Renal Failure (CRF); Graft Failure; Transplant; Failure, Kidney; Renal Transplant Rejection
Keywords: kidney transplantation; chronic renal failure; immunosuppressive therapy; elderly; pharmacokinetic; tacrolimus; everolimus; mycophenolate sodium; serious adverse events; biopsy; Cystatin C; metabolic effects; Left Ventricular Mass (LVM); Left Ventricle Ejection Fraction
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Everolimus; lactitol; Mycophenolic Acid; Prednisone; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): Number of patients: 45 Everolimus: initial dose of 1 mg BID. Doses will be adjusted in order to maintain Everolimus whole blood trough concentrations between 3-8 ng/ml.
  Tacrolimus: initial dose of 0.1 mg/kg/day. Doses will be adjusted in order to maintain Tacrolimus whole blood trough concentrations between 2- 4 ng/ml thereafter.
  Corticosteroids: as clinical practice.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — This is a 5-years prospective, randomized, exploratory, single-center, parallel group trial that includes renal transplanted elderly patients (≥ 60 years old) randomized between months 1 and 3 after transplantation to be maintained under MPS/TAC regimen or be switched to EVL/low-TAC.
  Everolimus: initial dose of 1 mg BID. Doses will be adjusted in order to maintain Everolimus whole blood trough concentrations between 3-8 ng/ml.
  Tacrolimus: initial dose of 0.1 mg/kg/day. Doses will be adjusted in order to maintain Tacrolimus whole blood trough concentrations between 2- 4 ng/ml thereafter.
  Corticosteroids: as clinical practice.
  Other Names: Certican (NOVARTIS); Myfortic (NOVARTIS); Prednisone (generic)

SUMMARY:
An exploratory study of the efficacy and safety of a regimen consisted of Everolimus plus low tacrolimus for the immunosuppression in renal transplantation in the elderly.

To evaluate the pharmacokinetics of immunosuppressants that have been little studied in this population.

To evaluate whether the polymorphism of the genes that determine the expression of metabolizing enzymes and transporters of xenobiotics interfere in the elderly, also in the younger population, absorption and metabolism of immunosuppressants.

To evaluate the potential minimization of immunosuppression in this population refers to how does the re-population of peripheral lymphocytes, in this age group, after the use of lymphocyte-depleting agents such as thymoglobulin and subsequently maintained with two regimes.

Clarify which markers of renal filtration exist today, cystatin C and serum creatinine, is the right to monitor renal function in elderly transplanted.

DETAILED DESCRIPTION:
Objectives: The objective of this study is to evaluate the safety and efficacy of everolimus (EVL) combined with low dose of Tacrolimus in comparison with Mycophenolate Sodium (MPS) combined with standard dose of Tacrolimus as immunosuppressive therapy for elderly recipients of kidney transplantation.

Comparison between the two study arms of:

Primary Objective:

1. Composite efficacy failure demonstrated by graft loss and/or death with functional graft and/or GFR (Glomerular Filtration Rate determined by EDTA-Cr51) < 50 ml/min at the end of first year after transplantation and every year until the fifth year.

Secondary Objectives:

1. Pharmacokinetic study of immunosuppressive drugs (Tacrolimus, Everolimus and Mycophenolate Sodium) in the study population at days 7, 30, 60, 67, 90 and 180 post-transplant.
2. Serious adverse events (as internationally defined by ICH-GCP) every year, for five years.
3. Biopsy proven acute rejection rated every year, for five years.
4. Identify which of the renal filtration markers existing today, Cystatin C or Serum Creatinine, is more adequate to monitor renal function in elderly transplant and to develop abbreviated equations for eGFR from day 7 on.
5. Evaluation of other metabolic effects (bone density at month 12 post-transplant; vitamin D at months 2 and 12 post-transplant; and gonadal function at months 1 and 12 post-transplant) and Quality of Life at months 1, 12, 18, 24, 36, 48 and 60 post-transplant in the study population.
6. Left Ventricular Mass (LVM) and Left Ventricle Ejection Fraction (LVEF) measured by echocardiography at the end of the first year.

ELIGIBILITY:
Inclusion Criteria:

* All renal (only) male and female recipients aged ≥ 60, years undergoing kidney transplantation from a living or deceased donor, including Expanded Criteria Donors (ECD).
* Panel Reactive Antibody (PRA) < 30%.
* Patients who consented to participate in the study by signing the informed consent form before the transplant surgery to the 1st post-operative day).

Exclusion Criteria:

* Allergy to any of proposed medications
* Patients with any active infection including HBV, HCV and HIV.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of functional graft | The study is planned to analyze all patients at the end of the fifth year after transplantation. However, an interim analysis will be done at the end of each year.
  Composite efficacy failure demonstrated by graft loss and/or death with functional graft and/or GFR (Glomerular Filtration Rate determined by EDTA-Cr51) < 50 ml/min at the end of first year after transplantation and every year until the fifth year.

SECONDARY OUTCOMES:
Pharmacokinetic of Tacrolimus | Days: 7, 30, 60, 67, 90, 180.
  Pharmacokinetic of Tacrolimus in the study population at days 7, 30, 60, 67, 90 and 180 post-transplant.
Serious adverse events | Every year, for five years
  Evaluate serious adverse events (as internationally defined by ICH-GCP).
Biopsy | Every year, for five years
  Biopsy proven acute rejection rated every year, for five years.
Renal filtration markers | Days: 7, 30, 37, 60, 67, 90, 180. Months: 12, 18, 24, 36, 48, 60
  Identify which of the renal filtration markers existing today, Cystatin C or Serum Creatinine, is more adequate to monitor renal function in elderly transplant and to develop abbreviated equations for eGFR from day 7 on.
Bone density | Month 12
  Evaluation of bone density at month 12 post-transplant.
Vitamin D | Months: 2, 12.
  Evaluation of vitamin D at months 2 and 12 post-transplant.
Gonadal function | Months: 1, 12.
  Evaluation of gonadal function at months 1 and 12 post-transplant.
Quality of Life | Months: 1, 12, 18, 24, 36, 48, 60.
  Evaluate Quality of Life at months 1, 12, 18, 24, 36, 48 and 60 post-transplant in the study population.
Left Ventricular Mass (LVM) | Month: 12.
  Left Ventricular Mass (LVM) measured by echocardiography at the end of the first year.
Left Ventricle Ejection Fraction (LVEF) | Month: 12.
  Left Ventricle Ejection Fraction (LVEF) measured by echocardiography at the end of the first year.
Pharmacokinetic of Everolimus | Days: 7, 30, 60, 67, 90, 180.
  Pharmacokinetic of Everolimus in the study population at days 7, 30, 60, 67, 90 and 180 post-transplant.
Pharmacokinetic of Mycophenolate Sodium | Days: 7, 30, 60, 67, 90, 180.
  Pharmacokinetic of Mycophenolate Sodium in the study population at days 7, 30, 60, 67, 90 and 180 post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Elias David-Neto, PhD, Principal Investigator — Clinical Hospital of the School of Medicine, University of Sao Paulo
Locations (1):
- Clinical Hospital of the School of Medicine, University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Romano P, Agena F, de Almeida Rezende Ebner P, Massakazu Sumita N, Kamada Triboni AH, Ramos F, Dos Santos Garcia M, Coelho Duarte NJ, Brambate Carvalhinho Lemos F, Zocoler Galante N, David-Neto E. Longitudinal Pharmacokinetics of Mycophenolic Acid in Elderly Renal Transplant Recipients Compared to a Younger Control Group: Data from the nEverOld Trial. Eur J Drug Metab Pharmacokinet. 2019 Apr;44(2):189-199. doi: 10.1007/s13318-018-0506-6. PMID 30229398